CLINICAL TRIAL: NCT06534385
Title: The Clean Air Study: High Efficiency Particulate Air (HEPA) Purifiers to Improve Indoor Air Quality and Health in Rural Alaska Homes
Brief Title: The Clean Air Study: HEPA Purifiers to Improve Indoor Air Quality and Health in Rural Alaska Homes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alaska Native Tribal Health Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1P20GM152302-01 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Air Pollution, Indoor
MeSH Terms: interventions — Air Filters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single group (Experimental): Participants receive HEPA purifiers and air monitoring equipment to operate daily for 12-weeks.
  Interventions: Device: Air purifier

INTERVENTIONS:
Device: Air purifier — Winix HEPA air purifier

SUMMARY:
Alaska Native children experience a high burden of respiratory disease, especially those in the Yukon-Kuskokwim (YK) Delta. Studies have shown that things like wood stove use, poor ventilation, and indoor tobacco smoke exposure can lead to poor indoor air quality inside the children's homes. This leads to more frequent and more severe respiratory infections in children.

In the Yukon-Kuskokwim (YK) Delta, it's common for homes to have exposure to woodstoves and tobacco use. Both of these activities affect indoor air quality in homes. We know that high efficiency particulate air (HEPA) purifiers can reduce particulate matter and make air quality better. One way that we measure air quality is through particulate matter (PM2.5). One of the few studies that looked at this in the YK Delta found that PM2.5 levels that were nearly twice as high as homes with woodstoves in other states. We believe it is important to reduce the PM2.5 in YK Delta homes. However, the few studies that looked at HEPA purifiers in rural Alaska did not include homes where smokers lived.

We know that breathing air with PM2.5 harms the lungs. We also know that HEPA filters can reduce PM2.5, which can mean reducing cough and wheeze in people with chronic lung conditions. We want to learn how HEPA filters work in homes with woodstoves or where a smoker lives, as it's likely these homes may have more PM2.5 than other homes. We expect that using HEPA filters will make the indoor air better and will mean decreased respiratory symptoms.

We plan to include 15 households with a child less than 5 years old in the family. Households that join will be asked to:

* Set up study equipment in their homes.
* Run the study equipment for 12 weeks and do a weekly report of child's respiratory symptoms by phone or text.
* Return the air-quality monitor equipment to the study team and keep the HEPA filters.

DETAILED DESCRIPTION:
When a child has a pulmonology visit, the nurse will give the family a study flyer and invite them to learn more about the study. Participants that complete the informed consent process will be asked to: set up study equipment in their homes, operate the study equipment and do a weekly report of the child's respiratory symptoms for 12 weeks, and return the air monitoring equipment to the study team.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native participants residing in homes where woodstoves are used for heat or a smoker resides in the home.

Exclusion Criteria:

* Plan to move homes during the study period.
* Using HEPA air purifiers (other than the ones provided by the study).

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Indoor particulate matter (PM2.5) concentrations | 12-weeks
  Mean weekly home indoor particulate matter (PM2.5) concentrations

SECONDARY OUTCOMES:
Reported symptom-free days | 12-weeks
  paired analysis of mean symptom-free days with no reported respiratory symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Yukon Kuskowkim Health Corporation, Bethel, Alaska, United States